CLINICAL TRIAL: NCT05822726
Title: The Combination of PSMA-PET/MRI and p2PSA in Early Diagnosis of Prostate Cancer
Brief Title: The Combination of PSMA-PET/MR and p2PSA in Early Diagnosis of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPMP-001
Record Dates: First submitted 2023-03-22; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; PSMA; p2PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combination of PSMA-PET/MR and p2PSA (Experimental)
  Interventions: Diagnostic Test: Prostate biopsy
- The combination of mpMRI and p2PSA (Active Comparator)
  Interventions: Diagnostic Test: Prostate biopsy

INTERVENTIONS:
Diagnostic Test: Prostate biopsy — Targeted guided puncture biopsy guided by B-ultrasound will be performed (in addition to 12-needle system biopsy, if PSMA-PET/MRI or mpMRI indicates a positive lesion, puncture biopsy should be added at the lesion displayed on image, the "12-needle system biopsy+X" scheme).

SUMMARY:
This is a single center prospective non-randomized controlled study.

The goal of this clinical trial is to figure out whether the combination of PSMA-PET/MR and PHI could add values to each method alone. The main questions it aims to answer are:

* Compare the diagnostic value of the combination with each alone and set up a diagnostic model.
* Compare the diagnostic value of PSMA-PET/MR+PHI to mpMRI+PHI.
* Evaluate the diagnostic value the combination of PHI and PSMA-PET/MR in suspected PCA patients.

Patients will experience mpMRI or PSMA-PET/MR and their blood samples will be used to test PSA and p2PSA. Prostate biopsy will be the golden standard.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative clinical judgment of suspected early prostate cancer (according to NCCN guidelines): meet PSA ≤ 20ng/ml and clinical stage<T3, while meeting one of the following criteria:

   ① Digital rectal examination revealed suspicious nodules of the prostate;

   ② Transrectal prostate ultrasound or MRI found suspicious lesions;

   ③ PSA>10 ng/ml；

   ④ PSA 4~10ng/ml, f/t PSA suspicious or PSAD value suspicious;
2. Aged between 18 and 85 years;
3. Generally in good health, able to tolerate and cooperate with research interventions, such as prostate biopsy and radical prostatectomy Etc;
4. Provide a signed and dated informed consent form;
5. Commit to complying with research procedures and cooperate in the implementation of the entire process of research.

Exclusion Criteria:

1. Preoperative clinical characteristics of suspected high-risk prostate cancer (according to NCCN guidelines): meet PSA>20 ng/ml or clinical stage ≥ T3;
2. Have received any treatment (endocrine therapy, radiotherapy, chemotherapy, prostate resection, etc.)
3. Have had prostatitis (infectious or non infectious) 3 months before the examination
4. Taking 5a reductase inhibitors
5. Previously diagnosed with prostate cancer
6. In the acute infection period and fever period;
7. Have a hypertensive crisis;
8. In the period of decompensation due to cardiac insufficiency;
9. Diseases with a tendency to severe bleeding;
10. In diabetes, blood sugar is unstable;
11. Have severe internal and external hemorrhoids, perianal or rectal lesions;
12. Combined with other systemic malignant tumors;
13. Implantation of functional electronic devices and various stimulators such as cardiac pacemakers, cochlear implants, and cardiac stents in vivo, with implants made of ferromagnetic materials (such as iron, cobalt, nickel, etc.);
14. A perfusion device implanted in the body, such as insulin or other perfusion pumps;
15. Have a history of surgery within the past 3 months, especially organ transplantation, heart and kidney surgery;
16. People with claustrophobia.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
biospy outcome | 12 months
  Compare the diagnostic value (including sensitivity, specificity, NPV and PPV) between both methods and set up a diagnostic model.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China